CLINICAL TRIAL: NCT05872763
Title: An Observational Cohort Study of Patients With Newly Diagnosed Unresectable Stage IIIB, IIIC, or IV Non-Small-Cell Lung Cancer (NSCLC) in China
Brief Title: A Study of Participants in China With Non-Small-Cell Lung Cancer That is Unable to be Treated With Surgery
Status: Active, not recruiting | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML44633
Record Dates: First submitted 2023-05-16; First posted 2023-05-24 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective cohort (Cohort 1): All cases of unresectable stage IIIB/IIIC/IV NSCLC newly diagnosed between January 2020 and the date of the study initiation will be collected. All these participants will be followed up until death or lost-to-follow-up or until 12 months after the last participant is enrolled in cohort 2 in the study.
- Prospective cohort (Cohort 2): The prospective enrollment of new cases of unresectable stage IIIB/IIIC/IV NSCLC will end up to 1 year after the first patient is enrolled (FPI) in Cohort 2.

SUMMARY:
This is a multicenter, observational cohort study in China with both primary prospective data collection and retrospective collection of prior treatment information from medical records, which enrolls and follows patients who are newly diagnosed with unresectable stage IIIB/IIIC/IV Non-Small-Cell Lung Cancer (NSCLC) in the selected sites.

This study aims to describe the clinical practice and long-term survival benefits of patients newly diagnosed with unresectable stage IIIB/IIIC/IV NSCLC. The study also seeks to explore the condition of biomarker tests utilization, and to assess potential economic impact on patients in the real world. The safety related events will also be summarized in this study.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1:

* Participants who have diagnosed with unresectable stage IIIB/IIIC/IV NSCLC
* Participants who have been diagnosed six months before the start of the study were required to have two complete tumor assessments within at least 6 months intervals after the diagnosis
* Participants who were newly diagnosed within six months before the start of the study were required to have complete baseline information (see section 6.4.1)
* Participants who have received standard first-line treatment defined by guideline CSCO (https://www.csco.org.cn/cn/index.aspx) and NCCN (https://www.nccn.org/)

Cohort 2:

* Participants who are newly diagnosed with unresectable Stage IIIB/IIIC/IV NSCLC after the start of the study
* Participants who are able to be followed up by the participating site
* Participants planned to receive first line anti-cancer treatment targeting unresectable stage IIIB/IIIC/IV NSCLC in the study site after study initiation

Exclusion Criteria:

* Participants who have received prior systematic treatment for unresectable Stage IIIB/IIIC/IV NSCLC
* Participants who have participated in any anti-cancer, regimen-specified clinical study of first-line treatment for unresectable Stage IIIB/IIIC/IV NSCLC

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will be conducted at multiple sites that will be selected from a pool of hospitals in China from 7 geographic regions (Northwest, Northeast, North, Southwest, South, Central, East) across China. And a target number of 7-10 sites across these regions were planned to be involved to ensure a relatively even number of patients to be enrolled from each region.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2023-08-11 (Actual); Primary Completion 2026-09-21 (Estimated); Study Completion 2026-09-21 (Estimated)

PRIMARY OUTCOMES:
Median Overall Survival (OS) | Up to 2 years
  OS is defined as the time from the date of the first administration of anti-cancer treatment until the date of death from any cause.
Median weeks on first-line treatment | Up to 2 years
  First-line treatment will be reported by class of treatment. Median, minimum, and maximum values will be used to summarize the number of weeks on the first line of treatment.

SECONDARY OUTCOMES:
Tumor Molecular Characteristics, measured by the presence of defined biomarkers | Up to 2 years
  The defined biomarkers to be identified are EGFR mutations, ALK rearrangement, ROS1 rearrangement, BRAF mutation, neurotrophic tyrosine receptor kinase [NTRK] gene fusion, KRAS mutations, and MET mutations. RET rearrangement, ERBB2 (HER2) mutation, and PD-L1 expression.
Treatment Cost to the Participant, measured by accrued fees; pharmacy fee, treatment fee, examinations fee, insurance coverage, and other medical costs | Up to 2 years
Number of participants with at least one adverse event, with severity determined according to National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0 (NCI-CTCAE v5.0) | Up to 2 years
Anti-cancer Treatment Duration | Up to 2 years
Number of Cycles of Anti-cancer Treatment | Up to 2 years
Number of Dose Modifications of Anti-Cancer Treatment | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (12):
- China (12):
  - Cancer Hospital Chinese Academy of Medical Sciences., Beijing
  - Beijing Chest Hospital, Beijing
  - Sichuan Provincial Cancer Hospital, Chengdu
  - Harbin Medical University Cancer Hospital, Harbin
  - Shandong Cancer Hospital, Jinan
  - Jiangsu Province Hospital (the First Affiliated Hospital With Nanjing Medical University), Nanjing
  - Guangxi Cancer Hospital of Guangxi Medical University, Nanning
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang
  - Shanxi Province Cancer Hospital, Taiyuan
  - Hubei Cancer Hospital, Wuhan
  - First Affiliated Hospital of Medical College of Xi'an Jiaotong University, Xi'an
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou

IPD SHARING:
Plan to Share IPD: No